CLINICAL TRIAL: NCT00944671
Title: A Single-Dose, Open-Label, Three-Period Crossover Study to Assess the Bioequivalence of Famotidine/Antacid Combination Tablets (FACT) Compared to Famotidine/Antacid EZ Chew Tablet Without Water and Famotidine/Antacid EZ Chew Tablet With Water
Brief Title: A Study to Assess the Bioequivalence of Famotidine/Antacid Combination Tablets Compared to Famotidine/Antacid EZ Chew Tablets (0208C-145)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0208C-145; 2009_622
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Results first posted 2015-06-24 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Heartburn
MeSH Terms: conditions — Heartburn | interventions — Famotidine; Calcium Carbonate; Magnesium Hydroxide; Water

ARMS (3):
- A (Active Comparator): Famotidine/antacid combination tablet with water
  Interventions: Drug: famotidine (+) calcium carbonate (+) magnesium hydroxide tablet
- B (Experimental): Famotidine/Antacid EZ Chew tablet without water
  Interventions: Drug: Comparator: famotidine (+) calcium carbonate (+) magnesium hydroxide EZ Chew tablet without water
- C (Experimental): Famotidine/Antacid EZ Chew tablet with water
  Interventions: Drug: Comparator: famotidine (+) calcium carbonate (+) magnesium hydroxide EZ Chew tablet with water

INTERVENTIONS:
Drug: famotidine (+) calcium carbonate (+) magnesium hydroxide tablet — A single dose of famotidine/antacid tablet with 120 mL of water in one of three treatment periods
  Arms: A
Drug: Comparator: famotidine (+) calcium carbonate (+) magnesium hydroxide EZ Chew tablet without water — A single dose of famotidine/antacid combination EZ Chew tablet without water in one of three treatment periods
  Arms: B
Drug: Comparator: famotidine (+) calcium carbonate (+) magnesium hydroxide EZ Chew tablet with water — A single dose of famotidine/antacid combination EZ Chew tablet with 120 mL of water in one of three treatment periods
  Arms: C

SUMMARY:
A study in 24 healthy subjects to assess the bioequivalence of Famotidine/Antacid EZ Chew tablet taken without water and with water compared to the Famotidine/Antacid tablet taken with water. Subjects will be given a single dose of each treatment separated by 5 to 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Female subject is not pregnant or lactating, Females of childbearing potential must use reliable means of contraception during the course of the study
* Subject is in good health
* Subject is able to abstain from smoking during the 24-hour periods before and during each treatment day

Exclusion Criteria:

* Subject has a history of stomach ulcers, other Gastrointestinal (GI) diseases or GI surgery
* Subject has a history of asthma or severe allergies to drugs or foods
* Subject currently uses prescribed or nonprescribed drugs on a regular basis
* Subject has a recent history of drug/alcohol abuse
* Subject consumes more than 6 cups of coffee per day
* Subject has unconventional or extreme dietary habits
* Subject has donated blood or has been in a clinical trial in which they received an investigational drug during the past 30 days
* Subject has a history of allergy or intolerance to antacids
* Female subject is known to be pregnant or is not using reliable means of contraception

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a single clinical research center in the US. Subjects were recruited via print advertisements and existing patient research files.
Pre-assignment Details: Prior to the first treatment period, Health Insurance Portability and Accountability Act (HIPAA) and informed consent were signed. For each subject a medical history was taken, physical examination and laboratory safety tests were conducted. No enrolled subjects were excluded from the trial before randomization.
Groups:
- Famotidine With Water/EZ Chew Without Water/EZ Chew With Water: Famotidine/antacid combination tablet with 120 mL of water, Famotidine/antacid combination EZ Chew tablet without water, Famotidine/antacid combination EZ Chew with 120 mL of water
- EZ Chew Without Water/EZ Chew With Water/Famotidine With Water: Famotidine/antacid combination EZ Chew tablet without water, Famotidine/antacid combination EZ Chew tablet with 120 mL of water, Famotidine/antacid combination tablet with 120 mL of water
- EZ Chew With Water/Famotidine With Water/EZ Chew Without Water: Famotidine/antacid combination EZ Chew tablet with 120 mL of water, Famotidine/antacid combination tablet with 120 mL of water, Famotidine/antacid combination EZ Chew tablet without water
- Famotidinewith Water/EZ Chew With Water/EZ Chew Without Water: Famotidine/antacid combination tablet with 120 mL of water, Famotidine/antacid combination EZ Chew tablet with 120 mL of water, Famotidine/antacid combination EZ Chew tablet without water
- EZ Chew Without Water/Famotidine With Water/EZ Chew With Water: Famotidine/antacid combination EZ Chew tablet without water, Famotidine/antacid combination tablet with 120 mL of water, Famotidine/antacid combination EZ Chew tablet with 120 mL of water
- EZ Chew With Water/EZ Chew Without Water/Famotidine With Water: Famotidine/antacid combination EZ Chew tablet with 120 mL of water, Famotidine/antacid combination EZ Chew tablet without water, Famotidine/antacid combination tablet with 120 mL of water
Period: Period I
Arm/Group | Famotidine With Water/EZ Chew Without Water/EZ Chew With Water | EZ Chew Without Water/EZ Chew With Water/Famotidine With Water | EZ Chew With Water/Famotidine With Water/EZ Chew Without Water | Famotidinewith Water/EZ Chew With Water/EZ Chew Without Water | EZ Chew Without Water/Famotidine With Water/EZ Chew With Water | EZ Chew With Water/EZ Chew Without Water/Famotidine With Water
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period II
Arm/Group | Famotidine With Water/EZ Chew Without Water/EZ Chew With Water | EZ Chew Without Water/EZ Chew With Water/Famotidine With Water | EZ Chew With Water/Famotidine With Water/EZ Chew Without Water | Famotidinewith Water/EZ Chew With Water/EZ Chew Without Water | EZ Chew Without Water/Famotidine With Water/EZ Chew With Water | EZ Chew With Water/EZ Chew Without Water/Famotidine With Water
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period III
Arm/Group | Famotidine With Water/EZ Chew Without Water/EZ Chew With Water | EZ Chew Without Water/EZ Chew With Water/Famotidine With Water | EZ Chew With Water/Famotidine With Water/EZ Chew Without Water | Famotidinewith Water/EZ Chew With Water/EZ Chew Without Water | EZ Chew Without Water/Famotidine With Water/EZ Chew With Water | EZ Chew With Water/EZ Chew Without Water/Famotidine With Water
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Famotidine With Water/EZ Chew Without Water/EZ Chew With Water | EZ Chew Without Water/EZ Chew With Water/Famotidine With Water | EZ Chew With Water/Famotidine With Water/EZ Chew Without Water | Famotidinewith Water/EZ Chew With Water/EZ Chew Without Water | EZ Chew Without Water/Famotidine With Water/EZ Chew With Water | EZ Chew With Water/EZ Chew Without Water/Famotidine With Water | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 24
Age, Continuous [Mean (Full Range); unit: years] | 29.8 [20 to 38] | 30.0 [20 to 45] | 29.8 [22 to 38] | 26.3 [22 to 38] | 30.8 [19 to 40] | 25.0 [20 to 39] | 28.6 [19 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 1 | 2 | 1 | 12
  Male | 2 | 1 | 1 | 3 | 2 | 3 | 12
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 1 | 1 | 2 | 1 | 2 | 2 | 9
  Caucasian | 3 | 3 | 2 | 2 | 2 | 2 | 14
  Native American | 0 | 0 | 0 | 1 | 0 | 0 | 1
Weight [Mean (Full Range); unit: Pounds] | 164.1 [151.5 to 186.1] | 152.2 [137.6 to 182.2] | 160.4 [148.5 to 175.2] | 164.8 [148.5 to 175.2] | 168.8 [132.7 to 200.0] | 165.3 [134.6 to 206.9] | 162.6 [132.7 to 206.9]

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC(0 to Infinity)) Following Single Dose Administration of Famotidine/Antacid Combination EZ Chew Without Water and Famotidine/Antacid Tablet With Water
Time Frame: Through 24 hours post-dose (½, 1, 1 ½, 2, 2 ½, 3, 4, 6, 8, 10, 12, 14, 24 hours post-dose)
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Famotidine/Antacid Combination EZ Chew Tablet Without Water | Famotidine/Antacid Combination Tablet With Water
Number analyzed (Participants) | 24 | 24
ng*hr/mL | 261.2 [227.9 to 299.3] | 248.0 [216.4 to 284.2]
Statistical Analysis 1: Comparison: Famotidine/Antacid Combination EZ Chew Tablet Without Water vs Famotidine/Antacid Combination Tablet With Water; Test type: Non-Inferiority or Equivalence — Given a 3-period crossover design, assuming a true within subject variance for natural log AUC of 0.029, 24 subjects completing the study, and alpha = 0.05, there is a 0.995 probability that the 90% confidence interval for the true geometric mean ratio of AUC for (famotidine antacid combination EZ Chew tablet without water/ famotidine antacid combination tablet with water) will be contained in (0.80, 1.25), given that the true ratio is one; Geometric Mean Ratio = 1.05, 90% CI [0.98 to 1.13]

2. Primary Outcome: Peak Plasma Concentration (Cmax) of Famotidine Following Single Dose Administration of Famotidine/Antacid Combination EZ Chew Without Water and Famotidine/Antacid Tablet With Water
Time Frame: Through 24 hours post-dose (½, 1, 1 ½, 2, 2 ½, 3, 4, 6, 8, 10, 12, 14, 24 hours post-dose)
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Famotidine/Antacid Combination EZ Chew Tablet Without Water | Famotidine/Antacid Combination Tablet With Water
Number analyzed (Participants) | 24 | 24
ng/mL | 45.5 [39.1 to 52.9] | 44.4 [38.1 to 51.7]
Statistical Analysis 1: Comparison: Famotidine/Antacid Combination EZ Chew Tablet Without Water vs Famotidine/Antacid Combination Tablet With Water; Test type: Non-Inferiority or Equivalence — Assuming a true within subject variance for natural log Cmax of 0.017, there is a 0.999 probability that the 90% confidence interval for the true geometric mean ratio of Cmax for (famotidine antacid combination EZ Chew tablet without water/ famotidine antacid combination tablet with water) will be contained in (0.80, 1.25), given that the true ratio is one; Geometric Mean Ratio = 1.03, 90% CI [0.93 to 1.13]

3. Secondary Outcome: Area Under the Curve (AUC(0 to Infinity)) Following Single Dose Administration of Famotidine/Antacid Combination EZ Chew With Water and Famotidine/Antacid Tablet With Water
Time Frame: Through 24 hours post-dose (½, 1, 1 ½, 2, 2 ½, 3, 4, 6, 8, 10, 12, 14, 24 hours post-dose)
Measure: Geometric Mean (95% Confidence Interval); unit: ng*h/mL
Arm/Group | Famotidine/Antacid Combination EZ Chew Tablet With Water | Famotidine/Antacid Combination Tablet With Water
Number analyzed (Participants) | 24 | 24
ng*h/mL | 260.1 [227.0 to 298.0] | 248.0 [216.4 to 284.2]
Statistical Analysis 1: Comparison: Famotidine/Antacid Combination EZ Chew Tablet With Water vs Famotidine/Antacid Combination Tablet With Water; Test type: Superiority or Other; Geometric Mean Ratio = 1.05, 90% CI [0.98 to 1.13]

4. Secondary Outcome: Peak Plasma Concentration (Cmax) of Famotidine Following Single Dose Administration of Famotidine/Antacid Combination EZ Chew With Water and Famotidine/Antacid Tablet With Water
Time Frame: Through 24 hours post-dose (½, 1, 1 ½, 2, 2 ½, 3, 4, 6, 8, 10, 12, 14, 24 hours post-dose)
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Famotidine/Antacid Combination EZ Chew Tablet With Water | Famotidine/Antacid Combination Tablet With Water
Number analyzed (Participants) | 24 | 24
ng/mL | 45.9 [39.4 to 53.4] | 44.4 [38.1 to 51.7]
Statistical Analysis 1: Comparison: Famotidine/Antacid Combination EZ Chew Tablet With Water vs Famotidine/Antacid Combination Tablet With Water; Test type: Superiority or Other; Geometric Mean Ratio = 1.03, 90% CI [0.93 to 1.14]

ADVERSE EVENTS:
Groups:
- Famotidine/Antacid Combination Tablet With Water: Famotidine/antacid combination tablet with 120 mL of water
- Famotidine/Antacid Combination EZ Chew Tablet Without Water: Famotidine/antacid combination EZ Chew tablet without water
- Famotidine/Antacid Combination EZ Chew Tablet With Water: Famotidine/antacid combination EZ Chew tablet with 120 mL of water
Arm/Group | Famotidine/Antacid Combination Tablet With Water | Famotidine/Antacid Combination EZ Chew Tablet Without Water | Famotidine/Antacid Combination EZ Chew Tablet With Water
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 3/24 | 4/24 | 5/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Famotidine/Antacid Combination Tablet With Water (N=24) | Famotidine/Antacid Combination EZ Chew Tablet Without Water (N=24) | Famotidine/Antacid Combination EZ Chew Tablet With Water (N=24)
Dysmenorrhea (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 4 (4)
Stomach discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope vasovagal (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.